CLINICAL TRIAL: NCT04865484
Title: Prospective Randomized Comparative Study of the Treatment of Multisegmental Fibrostenosing Crohn's Disease. Surgical Resection Plus Endoscopic Stricturotomy Versus Surgical Resection Plus Strictureplasty
Brief Title: Prospective Randomized Comparative Study of the Treatment of Multisegmental Fibrostenosing Crohn's Disease.
Acronym: SUREST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021ZSLYEC-020
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-03

CONDITIONS: Crohn Disease; Stricture; Bowel
MeSH Terms: conditions — Crohn Disease; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRES group (Experimental): Surgical resection plus endoscopic stricturotomy for multiple fibrous stenosis
  Interventions: Procedure: Surgical resection; Procedure: Endoscopic stricturotomy
- SRS group (Active Comparator): Surgical resection plus strictureplasty for multiple fibrous stenosis
  Interventions: Procedure: Surgical resection; Procedure: Strictureplasty

INTERVENTIONS:
Procedure: Surgical resection — Surgical resection of fibrostenotic area (>4cm)
Procedure: Endoscopic stricturotomy — Endoscopic stricturotomy of fibrostenotic area (≤4cm)
  Arms: SRES group
Procedure: Strictureplasty — Strictureplasty of fibrostenotic area (≤4cm)
  Arms: SRS group

SUMMARY:
Stenosis is one of the most frequent complications in patients with Crohn's disease (CD). In particular, CD patients with multi segmental intestinal strictures are often faced with short bowel syndrome after repeated or extensive surgical resection.

Strictureplasty conserves bowel and minimizes the risk of developing short-bowel syndrome in the short-term and, probably, long-term. Strictureplasty has become an established surgical option in the management of obstructive Crohn's disease, especially for multiple short fibrous strictures. It is particularly suitable for patients at risk for short-bowel syndrome.

Endoscopic management shows good efficacy and safety in the treatment of strictures in CD patients. The ECCO guideline recommended that endoscopic balloon dilatation is suitable to treat short [<5 cm] strictures of the terminal ileum in CD. Recently, Lan et al. reported that endoscopic stricturotomy appeared to be more effective in treating CD patients with anastomotic stricture than endoscopic balloon dilatation.

However, there is no scientific evidence for determining the most appropriate treatment for multiple fibrosis stenosis. We designed a prospective randomized comparative study of the treatment of multisegmental fibrostenosing Crohn's disease (surgical resection plus endoscopic stricturotomy versus surgical resection plus strictureplasty).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects had been diagnosed with CD for at least 3 months prior to screening, and the diagnosis of CD had clinical findings and endoscopic, imaging evidence, and was supported by histopathology reports
2. Subject is in remission from CD (CDAI score < 150)
3. Subjects had clinical findings of multiple fibrotic strictures of the bowel with obstruction (abdominal pain with distension, decreased stool frequency and / or symptoms of nausea and vomiting) and imaging evidence (MRE and bowel color ultrasound suggested intestinal fibrosis with greater than 50% reduction in diameter and greater than 20% thickening of the bowel wall with dilation of the proximal bowel), and endoscopic evidence (endoscopy was unable to pass)
4. Subjects had ≥ 2 small bowel strictures from duodenum to rectum and ≥ 20 cm maximum distance between coloanal and caudal strictures
5. Study process prior to initiation, the subject or subject's legal representative (if applicable) signed and dated a written informed consent form or any required documentation of privacy authorization
6. Female subjects who remained sexually and of childbearing potential with an ungerminated male partner, consented to adequate routine contraception throughout the study period starting with signing informed consent

Exclusion Criteria:

1. At the initial screening visit, subject presented with enterocutaneous fistula, abdominal abscess, evidence of gastrointestinal bleeding
2. Subjects were in active CD (CDAI score ≥ 150)
3. The subject had inflammatory activity in the stenotic bowel (as judged by a combination of blood inflammatory indices, endoscopy, ultrasound and imaging)
4. Presence of ileostomy, colostomy
5. Subjects had a history or evidence of adenomatous colonic polyps that had not been resected or had a history or evidence of dysplasia of the colonic mucosa, including low - or high-grade dysplasia, and an undiagnosed type of dysplasia
6. Subjects had suspected or confirmed ulcerative colitis, undiagnosed types of colitis, ischemic colitis, radiation enteritis, colitis associated diverticular disease, or microscopic colitis
7. Subjects had evidence of active infection during the screening period
8. Subject has active tuberculosis: chest X-ray performed within 3 months prior to week 0 results suggestive of suspected tuberculosis
9. Subjects with any defined inborn or acquired immunodeficiency (e.g., common various immunodeficiencies, human immunodeficiency virus [HIV] infection, organ transplantation)
10. Subjects had a clinically significant infection (e.g., pneumonia, pyelonephritis) or an ongoing chronic infection within 30 days prior to screening
11. The subject suffered from any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immune, endocrine / metabolic or other medical condition that, in the opinion of the investigator, would interfere with the outcome of the study or jeopardize the safety of the subject
12. The subject's medical history included malignancy
13. Subjects had abnormal laboratory results for any of the following during screening: hemoglobin < 5 g / dl; white blood cell (WBC) count < 3 × 10E9 / L; platelet count < 100 × 10E9 / L or > 1200 × 10E9 / L; alanine transaminase (ALT) or aspartate transaminase (AST) > 3 × upper limit of normal (ULN), and serum creatinine > 2 × ULN.
14. Subjects were unable to attend all study visits or comply with study flow plans female subjects were pregnant prior to study enrollment, during study enrollment, or plan to donate eggs during these time periods
15. Subjects were forced to consent to participate in the study
16. Investigators considered the subject unsuitable for endoscopic or surgical treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention-free survival | 52 weeks
  Percentage of patients who do not receive surgical or endoscopic intervention for obstruction recurrence

SECONDARY OUTCOMES:
Surgery-free survival | 52 weeks
  Percentage of patients who do not receive surgical intervention for obstruction recurrence
Obstructive score reduction | Week 4、12、20、28、36、44、52
  Obstructive score reduction compared to baseline
CDAI score reduction | Week 4、12、20、28、36、44、52
  CDAI score reduction compared to baseline
IBDQ score reduction | Week 4、12、20、28、36、44、52
  IBDQ score reduction compared to baseline
Adverse event rate | 52 weeks
  Percentage of adverse events
Total cost for intervention | 52 weeks
  Total cost for intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China